CLINICAL TRIAL: NCT05348083
Title: Bilateral Erector Spinae Plane Block (ESPB) Versus Posterior Quadratus Lumborum Block (p-QLB) for Postoperative Analgesia After Caesarean Section: an Observational Closed Mixed Cohort Study
Brief Title: Erector Spinae Plane Block (ESPB) Versus Quadratus Lumborum Block (QLB) for Postoperative Analgesia After Caesarean Section
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, ZANFINI BRUNO ANTONIO, Physician Anesthesiologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4412
Record Dates: First submitted 2021-12-15; First posted 2022-04-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Pain, Post Operative; Cesarean Section Complications; Anesthesia, Local; Obstetric Anesthesia Problems
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESPB: A prospective cohort of 25 patients ASA 2 (according to American Society of Anesthesiologists physical status classification) with normal singleton pregnancy, scheduled for elective caesarean section under spinal anesthesia without intrathecal morphine, who underwent bilateral echo-guided ESPB at T9 level at the end of surgery.
  Interventions: Procedure: ESPB
- p-QLB: A historical cohort of 25 patients ASA 2 (according to American Society of Anesthesiologists physical status classification) with normal singleton pregnancy, scheduled for elective caesarean section under spinal anesthesia without intrathecal morphine, who underwent bilateral echo-guided p-QLB at the end of surgery.

INTERVENTIONS:
Procedure: ESPB — Echo-guided bilateral ESPB performed at T9 level at the end of surgery with a mixture of ropivacaine 0.375% and epinephrine 5 mcg/mL 20 mL each side.
  Groups: ESPB

SUMMARY:
Management of pain after caesarean section represents an important anesthesiologic issue, since it is often suboptimal, leading to delayed functional recovery and chronic pain. Currently, the postoperative analgesic strategy mostly relies on intrathecal morphine (ITM) and multimodal analgesic regimen. Recently, the need for alterative opioid sparing techniques is emerging. Paraspinal fascial plane blocks, as quadratus lumborum block (QLB) and erector spinae plane block (ESPB) performed at T9 level, have therefore been proposed as alternatives to ITM, because of their demonstrated effect on visceral and somatic pain.

The aim of the study is to assess the efficacy, the feasibility and safety of bilateral ESPB compared to bilateral QLB for the management of postoperative pain after ceasarean section conducted under spinal anesthesia without ITM.

ELIGIBILITY:
Inclusion Criteria:

- Patients ASA 2 with normal singleton pregnancy, scheduled for elective caesarean section without intrathecal morphine, who underwent bilateral ESPB at the end of surgery an who gave informed consent to data collection.

Exclusion Criteria:

* Contraindications to spinal anesthesia;
* Contraindications to or a history of opioid dependence;
* Allergy to local anesthetics, acetaminophen, NSAIDs
* Inability to understand pain assessment scales or to use Patient Controlled Analgesia (PCA) pump;
* Patient refusal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is an observational comparative study, including a prospective cohort (the ESPB group) and a historical control group (the p-QLB group) from our institution.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption at 24 h | 24 hours from block performance
  Total morphine consumption at 24 hours from block performance

SECONDARY OUTCOMES:
Intensity of pain at time of block performance | Time of block performance, at the end of surgery
  NRS (Numeric Rating Scale) for pain at rest and on movement at time of block performance. NRS is an 11-point numeric scale ranging from 0 (= no pain) to 10 (=extreme pain)
Intensity of pain at 2 hours | 2 hours from block performance
  NRS (Numeric Rating Scale) for pain at rest and on movement at 2 hours from block performance. NRS is an 11-point numeric scale ranging from 0 (= no pain) to 10 (=extreme pain)
Intensity of pain at 6 hours | 6 hours from block performance
  NRS (Numeric Rating Scale) for pain at rest and on movement at 6 hours from block performance. NRS is an 11-point numeric scale ranging from 0 (= no pain) to 10 (=extreme pain)
Intensity of pain at 12 hours | 12 hours from block performance
  NRS (Numeric Rating Scale) for pain at rest and on movement at 12 hours from block performance. NRS is an 11-point numeric scale ranging from 0 (= no pain) to 10 (=extreme pain)
Intensity of pain at 24 hours | 24 hours from block performance
  NRS (Numeric Rating Scale) for pain at rest and on movement at 24 hours from block performance. NRS is an 11-point numeric scale ranging from 0 (= no pain) to 10 (=extreme pain)
Adverse events | Any time during the first 24 hours from block performance.
  Any adverse events, like sedation, itching, nausea, and other complications, particularly signs of local anesthetic toxicity, the occurrence or persistence of motor weakness at the lower extremities after spinal anesthesia recovery.
Time to first opioid request | Any time during the first 24 hours from block performance
  Interval time between block and first opioid analgesic request
Differences in hemodynamic parameters | Any time during the first 24 hours from block performance
  Any difference in hemodynamic parameters (non-invasive blood pressure, heart rate)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No